CLINICAL TRIAL: NCT05007418
Title: A Phase 1b, Open-Label Study of the Safety and Efficacy of Allogeneic Anti-CD38 A2 Dimeric Antigen Receptor (DAR)-T Cells in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study to Assess Allogeneic Anti-CD38 A2 Dimeric Antigen Receptor T Cells in Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 38DART-RRMM-101
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Anti-CD38 A2 DAR-T Cells; Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Intervention Model Description: To determine DLT and MTD, the design uses a 3+3 rule-based design. Dose escalation is permitted between successive cohorts based upon a specified algorithm, using discrete dosage steps.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-1492 (Experimental): Four dosing cohorts will be evaluated: Cohort 1 (1 × 10^5 donor DAR-T cells/kg); Cohort 2 (5 × 10^5 donor DAR-T cells/kg); Cohort 3 (1 × 10^6 donor DAR-T cells/kg); Cohort 4 (3 × 10^6 donor DAR-T cells/kg) where STI-1492 will be administered intravenously once.
  Interventions: Biological: STI-1492

INTERVENTIONS:
Biological: STI-1492 — Anti-CD38 A2 KOKI DAR T cells

SUMMARY:
This is a phase 1b, open-label, dose-escalation study of STI-1492 administered by a single intravenous infusion in subjects with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a phase 1b, open-label, multicenter, dose-escalation study of STI-1492 administered by a single intravenous infusion in subjects with relapsed or refractory multiple myeloma.

The study will determine the MTD and RP2D, assessing safety and preliminary efficacy using a conventional 3+3 study design with two design stages, an ascending dose stage followed by an expansion study.

Patients will be enrolled sequentially within each cohort and between cohorts during the dose escalation portion of the study with the staggered intervals of at least 28 days. Only one patient will be allowed to receive study treatment at any time through the end of the staggering period before the next subject may begin study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have relapsed or refractory multiple myeloma (RRMM) after having received prior lines of anti-myeloma treatments.
* Measurable disease as defined by one of the following: abnormal serum or M-protein levels; abnormal serum free light chain (FLC) assay; ≥ 30% clonal plasma cells in the bone marrow aspirate or biopsy sample
* Evidence of cell membrane CD38 expression as determined by immunohistochemistry (IHC) analysis ofbone marrow biopsy or extramedullary plasmacytoma
* Pulse oximetry ≥ 92% on room air
* Have a life expectancy ≥ 12 weeks
* Be willing and able to comply with the study schedule and all study requirements
* Willing to follow contraception guidelines

Exclusion Criteria:

* Previous treatment with any systemic therapy for multiple myeloma within 14 days prior to start of study dose
* Treatment with any cellular therapy within 8 weeks prior to start of study dose
* Have any unresolved toxicity ≥ Grade 2 from previous anticancer therapies
* A history of brain metastasis or spinal cord compression
* Has an ECOG performance status (PS) ≥ 3
* Has received allogeneic hematopoietic stem cell transplantation (HSCT) within 6 months, has active graft-versus-host disease (GvHD) following transplant, or is currently receiving immunosuppressive therapy following transplant
* Has any clinically significant low baseline lab results for hemoglobin, platelet counts, and neutrophil counts at screening unless resulting from underlying RRMM
* Has any clinically significant elevated baseline lab results for serum creatinine, AST or β2 microglobulin
* Abnormal INR or aPTT, unless on a stable dose of an anticoagulant
* Has known HIV or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C
* Is currently pregnant or breast feeding or planning on either during the study.
* Has an active bacterial, viral, or fungal infection
* Has active plasma cell leukemia
* Has extramedullary plasmacytoma(s)
* Has any significant medical condition, abnormality, or psychiatric illness that would prevent study participation
* Has left ventricular ejection fraction (LVEF) < 40%
* Has second primary malignancies (SPMs) in addition to multiple myeloma if the SPM has required therapy within the last 3 years or is not in complete remission
* Has any additional clinical history of the CNS or cardiovascular disease that would place the patient at an unacceptable risk if the patient participates in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety of STI-1492 | Baseline through study completion at up to approximately 54 months
  Safety as assessed by incidence of adverse events, SAEs, DLTs, neurotoxicity, cytokine release syndrome, host rejection, and laboratory abnormalities

SECONDARY OUTCOMES:
Overall response and duration | Baseline through study completion at up to approximately 54 months
  Response and duration according to the International Myeloma Working Group (IMWG) response criteria
Assessment of improvements in hypercalcemia, renal function, anemia and lytic bone lesions (CRAB criteria) | Baseline through study completion at up to approximately 54 months
  Assessment of improvement in CRAB criteria
Assessment of serum immunoglobulin levels | Baseline through study completion at up to approximately 54 months
  Assessment of serum immunoglobulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (3):
- United States (3):
  - UC Irvine, Orange, California
  - UC Davis, Sacramento, California
  - University of Oklahoma, Oklahoma City, Oklahoma